CLINICAL TRIAL: NCT06571461
Title: A Randomized, Open-label, Multi-center Phase III Clinical Study of Liposomal Irinotecan Combined With Oxaliplatin and S-1 Versus Gemcitabine Combined With Capecitabine for Postoperative Adjuvant Treatment of Pancreatic Cancer
Brief Title: Liposomal Irinotecan in Combination With Oxaliplatin and S-1 Versus Gemcitabine Combined With Capecitabine as Postoperative Adjuvant Therapy for Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE072-006
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — irinotecan sucrosofate; Oxaliplatin; S 1 (combination); Gemcitabine; Capecitabine

STUDY DESIGN:
Intervention Model Description: This study is designed as a phase III, two-arm, open-label, multi-center, randomized clinical trial comparing combination liposomal irinotecan, oxaliplatin and S-1 with gemcitabine + capecitabine when used as adjuvant therapy following resection for pancreatic ductal adenocarcinoma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NASOX：Liposomal Irinotecan; Oxaliplatin; S-1 (Experimental): Liposomal irinotecan at a dose of 50 mg/m² is administered intravenously over 90 minutes on D1. Oxaliplatin is administered at a dose of 60 mg/m² intravenously over 2 hours on D1. S-1 at a dose of 40 to 60mg twice daily is taken orally for 7 consecutive days, followed by a 7-day break. These medications are administered once every 2 weeks for a total of 12 cycles.
  Interventions: Drug: Liposomal Irinotecan; Drug: Oxaliplatin; Drug: S-1
- GX：Gemcitabine; Capecitabine (Active Comparator): Gemcitabine at a dose of 1000mg/m² is administered via intravenous infusion over 30 minutes on D1, 8, and 15 of a 28-day cycle. Capecitabine at a dose of 1660mg/m² per day in two divided oral doses is taken for 21 consecutive days, followed by a 7-day rest period. These medications are administered once every 4 weeks for a total of 6 cycles.
  Interventions: Drug: Gemcitabine; Drug: Capecitabine

INTERVENTIONS:
Drug: Liposomal Irinotecan — Liposomal Irinotecan：i.v. infusion
  Arms: NASOX：Liposomal Irinotecan; Oxaliplatin; S-1
Drug: Oxaliplatin — Oxaliplatin;：i.v. infusion
  Arms: NASOX：Liposomal Irinotecan; Oxaliplatin; S-1
Drug: S-1 — S-1: Oral
  Arms: NASOX：Liposomal Irinotecan; Oxaliplatin; S-1
Drug: Gemcitabine — Gemcitabine: i.v. infusion
  Arms: GX：Gemcitabine; Capecitabine
Drug: Capecitabine — Capecitabine: Oral
  Arms: GX：Gemcitabine; Capecitabine

SUMMARY:
This study will evaluate the efficacy and safety of adjuvant therapy with liposomal irinotecan in combination with oxaliplatin, and S-1 compared with capecitabine combined with capecitabine in participants with pancreatic ductal adenocarcinoma after radical surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients able and willing to provide a written informed consent aged 18-75 years.
2. Histologically confirmed resected ductal pancreatic adenocarcinoma (including adenosquamous carcinoma).
3. Undergone radical resection and confirmed macroscopic complete resection (R0 and R1).
4. Full recovery after surgery; able to start adjuvant treatment within 12 weeks after surgery.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
6. The main organs function well.

Exclusion Criteria:

1. Patients with other types of non-ductal tumor of the pancreas, including endocrine tumors or acinar cell adenocarcinoma, pancreatoblastoma, and solid-pseudopapillary tumor.
2. Macroscopic incomplete tumor removal (R2 resection).
3. Prior neo-adjuvant treatment, radiation therapy, or systemic therapy for pancreatic adenocarcinoma.
4. Presence or history of metastatic or locally recurrent pancreatic adenocarcinoma.
5. CA 19-9> 180 U / ml within 21 days before randomization.
6. The toxicity of previous therapy has not recovered to Grade 1 or below.
7. Known peripheral neuropathy (CTCAE ≥ Grade 2).
8. Known deficiency of dihydropyrimidine dehydrogenase (DPD)
9. Subjects with a confirmed diagnosis of Gilbert's syndrome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | Approximately 3 years.
  Disease-free survival is defined as the time from the date of randomization to the date of disease recurrence or death from any cause (whichever occurs first). Disease recurrence is defined as evidence of disease recurrence demonstrated by imaging assessment with CT or MRI scan and/or pathological diagnosis indicated by biopsy.

SECONDARY OUTCOMES:
Overall survival (OS) | Approximately 5 years.